CLINICAL TRIAL: NCT05493020
Title: The Association of Mukbang Watching Behavior and the Appetite of Children With Cancer Hospitalized for Radiotherapy and Chemotherapy: An Intensive Longitudinal Study
Brief Title: The Association Between Watching Mukbang Videos and the Appetite of Children With Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Other Study IDs: L2022SYSU-HL-089
Record Dates: First submitted 2022-07-27; First posted 2022-08-09 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Mukbang
Keywords: Mukbang; Childhood cancer; Appetite; Malnutrition; Quality of Life; Intensive Longitudinal Study
MeSH Terms: conditions — Neoplasms; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed children with cancer: Children with cancer who received at least one radiotherapy and chemotherapy during hospitalization
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — At baseline, the children's demographics, disease-related data, characteristics of "Mukbang"watching behavior, appetite, nutritional status, and quality of life data were collected. From the first day of radiotherapy or chemotherapy, 3 meals a day for 5 consecutive days were followed to track the children's appetite status and the characteristics of "Mukbang"watching behavior. Their nutritional status and quality of life were tracked at the end of treatment or when they were discharged from the hospital.

SUMMARY:
The purpose of this study is to record the "Mukbang" watching behavior and appetite of children with cancer during inpatient radiotherapy and chemotherapy through intensive longitudinal study, explore their correlation, and the impact on their nutritional status and quality of life, and formulate for clinical departments relevant interventions and management options provide a theoretical basis.

DETAILED DESCRIPTION:
World Health Organization（WHO） data shows that the prevalence of malnutrition in children with cancer is as high as 75%, which leads to decreased immune function in children with cancer, unsatisfactory treatment effect, increased adverse clinical outcomes, early tumor recurrence, prolonged recovery time, and death. risk factors such as increased rates. The "Global Childhood Oncology Initiative" proposed by WHO in 2020 pointed out that reducing hunger and malnutrition and improving the outcomes of children with cancer are one of the main tasks of providing best practices in pediatric oncology care.

The excessive consumption of the body caused by the cachexia of the tumor itself cannot be changed. Nutritional intake is the only adjustable factor for malnutrition in children with tumors. Loss of appetite is the main reason for insufficient nutritional intake. Numerous clinical studies have explored the nutritional management of children with cancer. However, most nutritional interventions are ineffective due to poor appetite and food intake in children.

The investigation in the clinical ward found that in order to cope with the problem of loss of appetite, many children with cancer took the initiative to watch "Mukbang" during hospitalization to relieve gastrointestinal symptoms and increase appetite. At present, studies have shown that "Mukbang" may have the potential to improve the appetite of children with tumors. In addition, watching "Mukbang" is a way that children actively choose to increase their appetite, which has better acceptability.

Intensive longitudinal study can explain the dynamic changes of children's behavior and appetite when watching "Mukbang" videos by sampling in a natural context for a short period of time and multiple times, and based on real-time data, further Explain in detail the persistent effect of watching "Mukbang" video behaviors on appetite.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-18；
* Children who conform to the Notice on Printing and Distributing the Diagnosis and Treatment Specifications for 12 Diseases Related to Hematological Diseases and Malignancies in Children (2021 Edition) issued by the General Office of the National Health and Health Commission;
* Experienced at least one complete cycle of chemotherapy and radiotherapy.

Exclusion Criteria:

* Children with severe cardiopulmonary disease, severe infection, severe organ damage, genetic metabolic disease, immunodeficiency disease or mental illness;
* Children with eye and ear dysfunction at the same time, resulting in the inability to watch and listen to videos.

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 178 children with cancer who have received at least one radiotherapy or chemotherapy during hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Appetite | Appetite change over 5 days during chemoradiotherapy from baseline
  The appetite will be assessed by Cancer Appetite and Symptom Questionnaire(CASQ) . The questionnaire consisted of 12 items, each item ranged from 0 to 4 points, and the total score of the questionnaire ranged from 0 to 48 points. The lower the total score, the worse the patient's appetite.
Mukbang Watching Features | Mukbang Watching Features change over 5 days during chemoradiotherapy from baseline
  The "Mukbang" watching features will be assessed by a questionnaire designed by the researcher and recorded by the subjects themselves, including watching time, watching rate, watching preferences and watching experience.

SECONDARY OUTCOMES:
Nutritional status | Change in nutritional status over 7 days from baseline
  The nutritional status will be assessed by using the Subjective Global Nutritional Assessment（SGNA）. Assessment included the children's recent height, weight, parental height, dietary intake, changes in appetite, frequency and duration of gastrointestinal symptoms, and recent physical activity and changes. This provides a comprehensive assessment of the nutritional status of children, with ratings classified as well-nourished, moderately malnourished or severely malnourished.
Quality of Life in children with cancer | Change in quality of life over 7 days from baseline
  The quality of life in children with cancer will be assessed by using the Pediatric Quality of Life Inventory Measurement Models 3.0（PedsQLTM-3.0-cancer）.The model has a total of 27 items, including 8 subscales, each item used a 5-point Likert scale, (0=never, 1=almost never, 2=sometimes, 3=often, 4 = almost always), higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No